CLINICAL TRIAL: NCT00453999
Title: Phase II, Multicenter, Randomized, Double-Mask, Double-Dummy Study Comparing Efficacy and Safety of Intravenous Peramivir Once Daily Versus Oral Oseltamivir Twice Daily in Adults With Acute Serious or Potentially Life-Threatening Influenza
Brief Title: Evaluation of Efficacy and Safety of Peramivir in Adults With Acute Serious or Potentially Life-threatening Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCX1812-201
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-01

CONDITIONS: Influenza
Keywords: influenza; flu
MeSH Terms: conditions — Influenza, Human | interventions — peramivir; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Peramivir 200 mg (Experimental): Peramivir 200 mg administered intravenously once daily for 5 days (5 doses)
  Interventions: Drug: Peramivir 200 mg
- Arm 2: Peramivir 400 mg (Experimental): Peramivir 400 mg administered intravenously once daily for 5 days (5 doses)
  Interventions: Drug: Peramivir 400 mg
- Arm 3: Oseltamivir (Experimental): Oseltamivir 75 mg oral suspension administered orally twice daily for 5 days (10 doses)
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Peramivir 200 mg — Peramivir (200 mg in 100 mL of solution) intravenous infusion (over 15 minutes) and an orally administered oseltamivir placebo suspension (6.25 mL) treatment
  Arms: Arm 1: Peramivir 200 mg
Drug: Peramivir 400 mg — Peramivir (400 mg in 100 mL of solution ) intravenous infusion (over 15 minutes) and an orally administered oseltamivir placebo suspension (6.25 ml)
  Arms: Arm 2: Peramivir 400 mg
Drug: Oseltamivir — Placebo peramivir infusion (over 15 minutes) and a 75-mg dose of oseltamivir suspension (6.25 mL)
  Arms: Arm 3: Oseltamivir

SUMMARY:
This study has been designed as a randomized, double-blind, controlled, study to evaluate the efficacy and safety of two once daily intravenous peramivir regimens (200 mg and 400 mg) versus oral oseltamivir phosphate (75 mg twice daily) in hospitalized subjects with acute serious or potentially life threatening influenza. Study treatments will be provided for up to 5 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age, male or female
* Able to provide informed consent, or for whom consent may be provided by guardian
* Presence of fever at time of screening of ≥38.0°C (≥ 100.0°F) taken orally, or ≥38.5°C (≥101.2°F) taken rectally. This requirement is waived if the subject has (1) a history of fever within 24 hours prior to screening and administered any antipyretic(s) in the 24 hours prior to screening, or (2) has no history of documented fever as defined above, but reports a symptom of feverishness at some time during 48 hours prior to screening
* Presence of at least 1 respiratory symptom (cough, sore throat, nasal congestion/symptoms) of any severity (mild, moderate, severe)
* Presence of at least 1 constitutional symptom (headache, myalgia, feverishness, malaise, fatigue) of any severity (mild, moderate, severe)
* Onset of illness no more than 72 hours before presentation. Time of onset of illness defined as either (1) the time when temperature (oral or rectal) was elevated (at least 1°C of elevation-oral temperature), OR (2) the time when the subject experienced the presence of at least 1 respiratory symptom AND the presence of at least 1 constitutional symptom
* Presence of 1 or more of the following factors in a subject willing to be hospitalized for inpatient observation and treatment:
* Age ≥60 years
* Presence of chronic obstructive pulmonary disease (COPD) or other chronic lung disease requiring daily pharmacotherapy
* History of congestive heart failure with or without medically significant recent change in cardiac status, but without signs or symptoms compatible with NYHA Class IV functional status
* Presence of diabetes mellitus, clinically stable or unstable
* Transcutaneous oxygen saturation <94% without supplemental oxygen for at least 5 minutes, or a medically significant decrease in oxygen saturation from an established baseline value
* Systolic blood pressure <90 mmHg
* Severity of illness that, in the Investigator's judgment, justifies hospitalization of the subject for supportive care
* Positive rapid antigen test (RAT) for influenza A and/or influenza B (using an approved test kit) or other test for influenza virus antigen performed in a clinical laboratory at the screening/enrollment evaluation
* Females of childbearing potential must report one of the following:
* Be surgically sterile or clinically post-menopausal
* Have been sexually abstinent 4 weeks prior to date of screening evaluation and be willing to remain abstinent through 4 weeks after study-drug administration for all perimenopausal women or women of child-bearing potential
* Use oral contraceptives or other form of hormonal birth control including hormonal vaginal rings or transdermal patches and have been using these for 3 months prior through 4 weeks after study-drug administration for all perimenopausal women or women of child-bearing potential
* Use an intra-uterine device (IUD), or adequate barrier contraception (or double-barrier method such as condom or diaphragm with spermicidal gel or foam) as birth control 4 weeks prior to date of screening evaluation through 4 weeks after study drug administration for all perimenopausal women or women of child-bearing potential

Exclusion Criteria:

* Immunized against influenza with live attenuated virus vaccine in the previous weeks
* Treatment with any dose(s) of rimantadine, amantadine, zanamivir, or oseltamivir in the previous 7 days
* Current clinical evidence of a recognized or suspected acute non-influenzal infectious illness with onset prior to Screening
* Serum creatinine laboratory result at Screening >1.6 mg/dL or a result >25% above the upper limit of normal for the laboratory performing the test
* History of clinically significant proteinuria (≥1000 mg/24 hrs)
* History of moderate or severe renal impairment and/or previous clinical laboratory data indicating an estimated creatinine clearance <50 mL/min during the previous 12 months
* Electrocardiogram (ECG) at Screening visit showing evidence of acute ischemia, or presence of a medically significant dysrhythmia
* Presence of cardiac signs or symptoms compatible with NYHA Class III or Class IV functional status for congestive heart failure or angina (see NYHA Appendix V)
* Presence of diagnosed COPD or other chronic lung condition requiring either continuous or intermittent oxygen therapy as an outpatient. Note: Subjects who are determined to require acute supplemental oxygen therapy at the time of Screening and/or at hospital admission may be enrolled, if exclusion criteria #13 or #14 are not applicable.
* History of organ transplantation during the previous 12 months
* Known HIV infection with most recent CD4+ T-cell count ≤350 cells/mL
* History of diagnosis of any type of cancer (hematologic or solid tumor), that has required chemotherapy or radiation therapy in the previous 12 months, excluding non-melanomatous localized skin cancer
* Presence of ongoing requirement for chronic mechanical ventilation, either via oral or nasotracheal intubation or via tracheostomy, or chronic or intermittent requirement for BiPAP (bilevel positive airway pressure) at screening. Note: Subjects who require intermittent CPAP treatment for sleep apnea (without oxygen supplementation) may be enrolled
* Subjects who require acute mechanical ventilatory support of any type at the time of screening.
* History of alcohol abuse or drug addiction during the previous 12 months
* Participation in a clinical study of an experimental medication or other treatment during the previous 4 weeks
* Previous treatment with intravenous or intramuscular peramivir
* Women who are pregnant (positive serum or urine pregnancy test), who are attempting to become pregnant, or who are breast-feeding
* Subjects who have been hospitalized due to a condition other than acute influenza and in whom influenza is diagnosed during hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (83):
- United States (41):
  - Pulmonary Associates of Mobile, P.C., Mobile, Alabama
  - St. Bernards Research Center/Clopton Clinic, Jonesboro, Arkansas
  - Pulmonary Consultants & Primary Care Physicians Medical Group, Inc., Orange, California
  - University of California Irvine Medical Center, Orange, California
  - University of California Davis Medical Center, Department of Emergency Medicine, Sacramento, California
  - Good Samaritan Hospital, San Jose, California
  - National Jewish Medical and Research Center, Clinical Research Unit, Denver, Colorado
  - Orlando Regional Healthcare, Orlando, Florida
  - James A. Haley Veterans Hospital, Department of Infectious Disease, Tampa, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Infectious Disease Specialists of Atlanta, P.C., Decatur, Georgia
  - St. Joseph's/Candler Health System, Inc., Savannah, Georgia
  - Idaho Falls Infectious Diseases, PLLC, Idaho Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Springfield Clinic, LLP, Springfield, Illinois
  - Wishard Hospital/Indiana University, Indianapolis, Indiana
  - Infectious Disease of Indiana, PSC, Indianapolis, Indiana
  - Natchitoches Internal Medicine, Natchitoches, Louisiana
  - Louisiana State University Health Sciences Center-Shreveport, Shreveport, Louisiana
  - VA Maryland Health Care System, Baltimore, Maryland
  - Franklin Square Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University School of Medicine, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - William Beaumont Hospital Troy, Troy, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Hackensack University Medical Center, Department of Infectious Disease, Hackensack, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Rochester General Hospital/University of Rochester, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Lowcountry Infectious Diseases, P.A., Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Veterans Affairs Medical Center, Salem, Virginia
  - Franciscan Health System, Tacoma, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - Prince Of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Cairns Base Hospital, Cairns, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Gold Coast Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Repatriation General Hospital, Daw Park, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Canada (10):
  - Kelowna General Hospital, Kelowna, British Columbia
  - Hamilton Health Sciences-McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton-L424, Hamilton, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Mount Sinai Hospital / Toronto Medical Laboratories, Toronto, Ontario
  - Center de Sante et des Services Sociaux de Chicoutimi, Chicoutimi, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec-Pavillon CHUL, Québec, Quebec
  - Centre de sante et de services sociaux Rimouski-Neigette (CSSSRN), Rimouski, Quebec
  - Division of Infectious Diseases, Saskatoon, Saskatchewan
- Hong Kong (4):
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - United Christian Hospital, Hong Kong
  - The Prince of Wales Hospital, Shatin - New Territories
- New Zealand (3):
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Tauranga Hospital, Tauranga
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Africa (14):
  - Global Clinical Trial Center, Port Elizabeth, E. Cape
  - Genclin Corporation, Bloemfontein, Free State
  - Benmed / Pentagon Hospital, Benoni, Gauteng
  - Private Practice, Cape Town, Gauteng
  - Newgate Centre, Johannesburg, Gauteng
  - DJW Navorsing, Krugersdorp, Gauteng
  - Medforum Hospital, Pretoria, Gauteng
  - Eugene Marais Hospital, Pretoria, Gauteng
  - Global Clinical Trials (GCT), Pretoria, Gauteng
  - Dr Bhorat, Soweto, Gauteng
  - Sebastian, P, Durban, KZ-Natal
  - Eksteen, MC, Mbombela, Mpumalanga
  - Dr. L.J. van Zyl, Worcester, W Cape
  - N1 City Hospital, Cape Town, WC

REFERENCES:
- [Derived] Ison MG, Hui DS, Clezy K, O'Neil BJ, Flynt A, Collis PJ, Simon TJ, Alexander WJ. A clinical trial of intravenous peramivir compared with oral oseltamivir for the treatment of seasonal influenza in hospitalized adults. Antivir Ther. 2013;18(5):651-61. doi: 10.3851/IMP2442. Epub 2012 Oct 30. PMID 23111657

RESULTS

PARTICIPANT FLOW:
Groups:
- Peramivir 400 mg: Peramivir (400 mg in 100 mL of solution) intravenous infusion (over 15 minutes) and an orally administered oseltamivir placebo suspension (6.25 mL)
Period: Overall Study
Arm/Group | Peramivir 200 mg | Peramivir 400 mg | Oseltamivir
Started | 45 | 46 | 46
Completed | 40 | 41 | 43
Not Completed | 5 | 5 | 3
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Subject Request | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Peramivir 200 mg | Peramivir 400 mg | Oseltamivir | Total
Number analyzed (Participants) | 45 | 46 | 46 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (24.0) | 58.5 (20.9) | 62.0 (21.3) | 59.2 (22.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 25 | 76
  Male | 20 | 20 | 21 | 61
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 23 | 21 | 20 | 64
  Black or African American | 8 | 14 | 12 | 34
  Asian | 13 | 10 | 13 | 36
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Other | 0 | 1 | 1 | 2
Height [Mean (Standard Deviation); unit: cm] | 163.0 (9.9) | 161.6 (11.8) | 168.4 (11.8) | 164.4 (11.5)
Weight [Mean (Standard Deviation); unit: kg] | 64.9 (19.8) | 72.4 (22.9) | 79.5 (22.7) | 72.4 (22.5)
Duration of Illness at Randomization [Number; unit: participants]
  < 48 hours | 31 | 32 | 31 | 94
  >= 48 hours to <=72 hours | 14 | 14 | 15 | 43
Initial Composite Symptom Score [Mean (Standard Deviation); unit: units on a scale] — Initial Composite Symptom Score is defined as the sum of the 7 symptoms of influenza recorded at the predose visit. (cough; sore throat; nasal congestion; myalgia [aches and pains]; headache; feverishness; and fatigue), each graded on a 4-point severity scale (0, absent; 1, mild; 2, moderate; 3, severe); for the composite score, individual scores were summed, with a range from 0 to 21. Data were available for 122 participants (39 in the Peramivir 200 mg group; 41 in the Peramivir 400 mg group; and 42 in the Oseltamivir group).
  units on a scale | 12.7 (5.19) | 12.2 (5.95) | 12.3 (5.46) | 12.4 (5.51)
Current Smoking Status [Number; unit: participants] — A smoker was defined as a subject who had smoked cigarettes in the last 30 days or currently used other tobacco products. Data were available for 135 participants (44 in the Peramivir 200 mg group; 45 in the Peramivir 400 mg group; and 46 in the Oseltamivir group).
  participants
    Smoker | 8 | 5 | 4 | 17
    Nonsmoker | 36 | 40 | 42 | 118
    Missing | 1 | 1 | 0 | 2
Influenza Infection [Number; unit: participants] — "Confirmed" included all subjects with confirmed influenza defined as a positive polymerase chain reaction (PCR) assay, positive viral culture, or paired serology showing a ≥ 4-fold increase in antibody to influenza A or B.
  participants
    Confirmed Influenza A | 26 | 34 | 30 | 90
    Confirmed Influenza B | 15 | 6 | 11 | 32
    Not confirmed | 4 | 6 | 5 | 15
Transcutaneous Oxygen Saturation at Randomization [Number; unit: participants]
  < 94% | 14 | 14 | 14 | 42
  >= 94% | 31 | 32 | 32 | 95

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinical Stability (Kaplan-Meier Estimate)
Description: Time to clinical stability was summarized overall and for individual clinical signs for each treatment group using the method of Kaplan Meier. Subjects who did not experience clinical stability were censored at the date of their last non-missing assessment during the study (whether this assessment occurred as an inpatient or as an outpatient).
Time Frame: 14 days
Population: The intent-to-treat infected (ITTI) population included all subjects who were randomized, received at least 1 dose of study drug, and had confirmed influenza infection by viral culture, PCR, and/or paired acute and convalescent serology specimens that demonstrated at least a 4-fold increase in antibody titer against influenza A or B.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Peramivir 200 mg | Peramivir 400 mg | Oseltamivir
Number analyzed (Participants) | 41 | 40 | 41
hours | 23.7 [16.0 to 38.9] | 37.0 [22.0 to 48.7] | 28.1 [22.0 to 37.0]
Statistical Analysis 1: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Test type: Superiority or Other; p = 0.306, Log Rank; Differences between groups by log-rank statistic stratified by oxygen saturation and duration of illness at randomization, and flu season

2. Secondary Outcome: Change From Baseline in Scores of Symptoms of Influenza
Description: Descriptive statistics for the change from baseline in each of the 7 symptoms of influenza (cough; sore throat; nasal congestion; myalgia [aches and pains]; headache; feverishness; and fatigue, each graded on a 4-point severity scale [0, absent; 1, mild; 2, moderate; 3, severe]) were tabulated by treatment group. Missing data were excluded.
Time Frame: Baseline, Days 2, 3, 4, 5, 10, and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peramivir 200 mg | Peramivir 400 mg | Oseltamivir
Number analyzed (Participants) | 41 | 40 | 41
units on a scale
  Sore Throat: Baseline | 1.3 (1.09) | 1.1 (1.17) | 1.2 (1.19)
  Sore Throat: Change at Day 2 | -0.2 (0.95) | -0.3 (1.09) | -0.3 (0.80)
  Sore Throat: Change at Day 3 | -0.8 (1.05) | -0.7 (1.24) | -0.8 (1.04)
  Sore Throat: Change at Day 4 | -0.9 (1.13) | -0.9 (1.24) | -1.1 (1.18)
  Sore Throat: Change at Day 5 | -1.1 (1.07) | -0.9 (1.20) | -1.1 (1.24)
  Sore Throat: Change at Day 10 | -1.2 (1.03) | -1.1 (1.15) | -1.2 (1.18)
  Sore Throat: Change at Day 14 | -1.2 (1.05) | -1.1 (1.16) | -1.1 (1.17)
  Nasal Congestion: Baseline | 1.3 (1.17) | 1.5 (1.03) | 1.3 (1.08)
  Nasal Congestion: Change at Day 2 | -0.2 (1.06) | -0.5 (0.82) | -0.3 (0.82)
  Nasal Congestion: Change at Day 3 | -0.7 (1.18) | -0.9 (0.99) | -0.8 (0.96)
  Nasal Congestion: Change at Day 4 | -0.8 (1.32) | -1.1 (1.06) | -1.0 (1.16)
  Nasal Congestion: Change at Day 5 | -0.9 (1.27) | -1.2 (1.17) | -1.1 (1.10)
  Nasal Congestion: Change at Day 10 | -1.1 (1.23) | -1.2 (1.27) | -1.1 (1.17)
  Nasal Congestion: Change at Day 14 | -1.0 (1.22) | -1.2 (1.17) | -1.3 (1.08)
  Cough: Baseline | 2.2 (0.73) | 2.0 (0.77) | 2.1 (0.76)
  Cough: Change at Day 2 | -0.4 (0.88) | -0.3 (0.74) | -0.2 (0.81)
  Cough: Change at Day 3 | -0.9 (0.91) | -0.9 (1.07) | -0.9 (0.87)
  Cough: Change at Day 4 | -1.1 (1.10) | -1.1 (1.05) | -1.0 (1.07)
  Cough: Change at Day 5 | -1.2 (0.97) | -1.1 (1.23) | -1.1 (1.17)
  Cough: Change at Day 10 | -1.4 (0.97) | -1.2 (1.07) | -1.3 (1.11)
  Cough: Change at Day 14 | -1.6 (1.06) | -1.4 (1.01) | -1.5 (1.09)
  Aches and Pains: Baseline | 1.8 (1.30) | 1.9 (1.13) | 1.9 (1.09)
  Aches and Pains: Change at Day 2 | -0.8 (1.01) | -0.8 (0.91) | -0.8 (1.08)
  Aches and Pains: Change at Day 3 | -1.3 (1.14) | -1.4 (1.18) | -1.4 (1.14)
  Aches and Pains: Change at Day 4 | -1.5 (1.28) | -1.6 (1.21) | -1.6 (1.21)
  Aches and Pains: Change at Day 5 | -1.6 (1.31) | -1.6 (1.23) | -1.7 (1.31)
  Aches and Pains: Change at Day 10 | -1.7 (1.38) | -1.7 (1.12) | -1.9 (1.09)
  Aches and Pains: Change at Day 14 | -1.7 (1.35) | -1.6 (1.11) | -1.7 (1.30)
  Fatigue: Baseline | 2.3 (0.78) | 2.0 (0.96) | 2.3 (0.82)
  Fatigue: Change at Day 2 | -0.9 (0.96) | -0.5 (1.12) | -1.0 (1.11)
  Fatigue: Change at Day 3 | -1.2 (1.02) | -1.0 (1.26) | -1.1 (1.17)
  Fatigue: Change at Day 4 | -1.4 (1.21) | -1.2 (1.30) | -1.6 (1.11)
  Fatigue: Change at Day 5 | -1.6 (1.09) | -1.3 (1.27) | -1.7 (1.09)
  Fatigue: Change at Day 10 | -1.7 (1.05) | -1.4 (1.13) | -1.7 (1.09)
  Fatigue: Change at Day 14 | -1.7 (1.13) | -1.6 (1.01) | -2.0 (0.97)
  Headache: Baseline | 1.5 (1.22) | 1.3 (1.34) | 1.4 (1.30)
  Headache: Change at Day 2 | -0.5 (1.11) | -0.5 (1.12) | -0.6 (0.94)
  Headache: Change at Day 3 | -0.9 (1.16) | -1.0 (1.26) | -1.0 (1.10)
  Headache: Change at Day 4 | -1.0 (1.25) | -1.1 (1.30) | -1.1 (1.30)
  Headache: Change at Day 5 | -1.2 (1.21) | -1.1 (1.28) | -1.3 (1.30)
  Headache: Change at Day 10 | -1.3 (1.24) | -1.2 (1.35) | -1.4 (1.26)
  Headache: Change at Day 14 | -1.3 (1.19) | -1.2 (1.35) | -1.3 (1.34)
  Feeling Feverish: Baseline | 2.1 (1.04) | 1.9 (0.99) | 1.8 (1.20)
  Feeling Feverish: Change at Day 2 | -1.4 (1.02) | -1.0 (0.94) | -1.0 (1.15)
  Feeling Feverish: Change at Day 3 | -1.5 (1.01) | -1.5 (0.93) | -1.6 (1.20)
  Feeling Feverish: Change at Day 4 | -1.8 (1.15) | -1.8 (0.97) | -1.6 (1.48)
  Feeling Feverish: Change at Day 5 | -1.9 (1.02) | -1.8 (1.02) | -1.8 (1.20)
  Feeling Feverish: Change at Day 10 | -2.0 (1.07) | -1.8 (1.00) | -1.8 (1.18)
  Feeling Feverish: Change at Day 14 | -1.9 (1.21) | -1.7 (1.01) | -1.8 (1.23)
Statistical Analysis 1: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Sore Throat: change from Baseline at Days 2, 3, 4, 5, 10, 14; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Nasal Congestion: change from Baseline at Days 2, 3, 4, 5, 10, 14; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Cough: change from Baseline at Days 2, 3, 4, 5, 10, 14; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Aches and Pains: change from Baseline at Days 2, 3, 4, 5, 10, 14; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Fatigue: change from Baseline at Days 2, 3, 4, 5, 10, 14; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Headache: change from Baseline at Days 2, 3, 4, 5, 10, 14; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Feeling Feverish: change from Baseline at Days 2, 3, 4, 5, 10, 14; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test

3. Secondary Outcome: Time to Resumption of Ability to Perform Usual Activities (Kaplan-Meier Estimate)
Description: Changes in each subject's ability to perform usual activities as determined from the visual analog scale (0 to 10, where 0 indicated subject was unable to perform usual activities at all and 10 indicated subject was able to perform all usual activities fully) were summarized by study visit and treatment group. The time to resumption of a subject's ability to perform usual activities was estimated using the method of Kaplan Meier. Subjects who did not return to the pre-study level of performance of usual activities were censored at the time of their last assessment. (Note: N is the number of ITTI participants with available data).
Time Frame: 14 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Peramivir 200 mg | Peramivir 400 mg | Oseltamivir
Number analyzed (Participants) | 40 | 39 | 41
hours | 8.8 [4.0 to 14.5] | 9.0 [6.8 to NA] — The number of observed events was too small to allow estimation of the required parameter. | 13.7 [10.0 to 20.7]
Statistical Analysis 1: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Test type: Superiority or Other; p = 0.276, Log Rank

4. Secondary Outcome: Incidence of Clinical Relapse of Influenza After Treatment (Number of Participants Experiencing Relapse During the Study)
Description: The number of subjects with clinical relapse, defined as changes in 2 or more signs of clinical stability to values outside the range of normalization criteria for a duration of at least 12 consecutive hours after clinical stability had been attained, were summarized by treatment group.
Time Frame: 14 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Peramivir 200 mg | Peramivir 400 mg | Oseltamivir
Number analyzed (Participants) | 41 | 40 | 41
participants | 0 | 0 | 0

5. Secondary Outcome: Time to Hospital Discharge (Kaplan-Meier Estimate)
Description: Time to discharge from hospital was estimated using the method of Kaplan Meier. Subjects who were not discharged from the hospital were censored at the time of their last assessment.
Time Frame: 14 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Peramivir 200 mg | Peramivir 400 mg | Oseltamivir
Number analyzed (Participants) | 41 | 40 | 41
hours | 4.0 [3.0 to 4.7] | 3.8 [2.7 to 4.8] | 4.0 [2.9 to 4.6]
Statistical Analysis 1: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Test type: Superiority or Other; p = 0.994, Log Rank

6. Secondary Outcome: Change in Amount of Influenza Virus in Nose and Throat (Influenza A and B Combined)
Description: Reduction in viral shedding, assessed as the change in quantitative viral titers and defined as the time-weighted change from baseline in TCID50/mL, was summarized for each treatment group.
Time Frame: Baseline, and 12, 24, 36, 48, 72, and 96 hours
Population: Among the 122 subjects with confirmed influenza (intent-to-treat infected [ITTI]) population, a total of 112 subjects had positive virus cultures obtained from baseline nasopharyngeal specimens.
Measure: Mean (Standard Deviation); unit: log10 TCID50/mL
Arm/Group | Peramivir 200 mg | Peramivir 400 mg | Oseltamivir
Number analyzed (Participants) | 39 | 34 | 39
log10 TCID50/mL
  Duration <48 Hours: Baseline | 3.6 (1.33) | 3.5 (1.01) | 3.4 (1.44)
  Duration <48 Hours: Change at 12 hours | -1.5 (1.33) | -1.6 (1.29) | -1.5 (1.01)
  Duration <48 Hours: Change at 24 hours | -2.5 (0.93) | -2.2 (0.84) | -2.2 (0.99)
  Duration <48 Hours: Change at 48 hours | -2.4 (0.93) | -2.9 (0.77) | -2.5 (1.45)
  Duration <48 Hours: Change at 96 hours | -2.8 (1.28) | -3.0 (0.97) | -2.8 (1.05)
  Duration ≥48 and ≤72 hours: Baseline | 2.8 (1.38) | 2.6 (1.35) | 2.5 (1.27)
  Duration ≥48 and ≤72 hours: Change at 12 hours | -1.1 (1.03) | -1.5 (1.27) | -0.7 (1.12)
  Duration ≥48 and ≤72 hours: Change at 24 hours | -1.4 (0.92) | -1.7 (1.22) | -1.0 (0.75)
  Duration ≥48 and ≤72 hours: Change at 48 hours | -1.8 (1.17) | -1.9 (1.16) | -1.5 (0.85)
  Duration ≥48 and ≤72 hours: Change at 96 hours | -2.6 (1.29) | -2.0 (1.38) | -1.7 (1.44)
Statistical Analysis 1: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Change from Baseline at 12 hours; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Change from Baseline at 24 hours; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Change from Baseline at 36 hours; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Change from Baseline at 48 hours; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Change from Baseline at 72 hours; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Peramivir 200 mg vs Peramivir 400 mg vs Oseltamivir; Change from Baseline at 96 hours; Test type: Superiority or Other; p > 0.05, Wilcoxon Rank Sum Test

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study drug administration through the follow-up period ending on Day 14.
Description: For subjects who experienced the same coded event more than once, only one event is presented.
Arm/Group | Peramivir 200 mg | Peramivir 400 mg | Oseltamivir
Serious Adverse Events (participants affected / at risk) | 2/45 | 8/46 | 4/46
Other Adverse Events (participants affected / at risk) | 25/45 | 21/46 | 19/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peramivir 200 mg (N=45) | Peramivir 400 mg (N=46) | Oseltamivir (N=46)
Pneumonia (Infections and infestations) | 0 | 3 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Viral myocarditis (Infections and infestations) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peramivir 200 mg (N=45) | Peramivir 400 mg (N=46) | Oseltamivir (N=46)
Diarrhoea (Gastrointestinal disorders) | 5 | 7 | 1
Nausea (Gastrointestinal disorders) | 2 | 5 | 4
Constipation (Gastrointestinal disorders) | 3 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0
Gingival Pain (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 4 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 2 | 0
Blood Alkaline Phosphatase Decreased (Investigations) | 0 | 0 | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 1
Blood Magnesium Decreased (Investigations) | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 1 | 0
Brain Natriuretic Peptide Increased (Investigations) | 0 | 1 | 0
Electrocardiogram Change (Investigations) | 1 | 0 | 0
Electrocardiogram Qt Prolonged (Investigations) | 1 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 1 | 0 | 0
Weight Decreased (Investigations) | 1 | 0 | 0
White Blood Cell Count Increased (Investigations) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Mood Altered (Psychiatric disorders) | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchial Secretion Retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 1 | 0
Bronchiectasis (Infections and infestations) | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 1
Fungal Skin Infection (Infections and infestations) | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Staphylococcal Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1
Dizziness Postural (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 2
Chest Pain (General disorders) | 1 | 0 | 0
Infusion Site Pain (General disorders) | 0 | 1 | 0
Infusion Site Pruritus (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Non-cardiac Chest Pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Vessel Puncture Site Haematoma (General disorders) | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 1
Vision Blurred (Eye disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No